CLINICAL TRIAL: NCT06941155
Title: A Randomized Controlled Trial on the Effects of Mobile-Based Gamified Combined Cognitive Bias Modification on OCD Symptoms, Obsessive Beliefs, Cognitive Biases, Depressive Symptoms and Distress in Adults Diagnosed With OCD
Brief Title: Gamified Combined Cognitive Bias Modification in Adults Diagnosed With OCD: Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Sıla Derin, PhD, Cilinical Psychologist, PhD, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 223S390
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Obsessive Compulsive Disorder (OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel groups: (1) gamified cognitive bias modification-combined (CBM-C), (2) standard CBM-C, or (3) placebo control. Each group will receive only one type of intervention throughout the study period. Interventions will be delivered independently and simultaneously via mobile phone, and there will be no crossover between conditions.
Who Masked: Participant
Masking Description: The participants will know that they will receive a treatment, but they will be blinded to randomization, i.e. will not know which groups they can be randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gamified-Combined Cognitive Bias Modification (Experimental): Participants in this group will receive the gamified version of the combined cognitive bias modification (CBM-C) intervention, consisting of eight sessions over four weeks (two sessions per week), delivered via mobile phone. The intervention includes both attention and interpretation bias modification tasks enhanced with gamification elements.
  Interventions: Behavioral: Gamified-Combined Cognitive Bias Modification
- Standart Combined Cognitive Bias Modification (Active Comparator): Participants in this group will receive the standard version of the combined cognitive bias modification (CBM-C) intervention, consisting of eight sessions over four weeks (two sessions per week), delivered via mobile phone. The intervention includes both attention and interpretation bias modification tasks, without any gamification features.
  Interventions: Behavioral: Standard Combined Cognitive Bias Modification
- Placebo Control (Placebo Comparator): Participants in this group will receive a placebo version of the standard combined cognitive bias modification (CBM-C) intervention, consisting of eight sessions over four weeks (two sessions per week), delivered via mobile phone. The placebo version retains the structure of the standard intervention but does not include any active bias modification components.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Gamified-Combined Cognitive Bias Modification — A gamified version of the combined cognitive bias modification (CBM-C) intervention, which includes both attention and interpretation bias modification tasks. The attention component is a modified dot-probe task, and the interpretation component consists of OCD-related scenarios with word-completion exercises. Gamification elements such as feedback and visual rewards are embedded to enhance motivation and engagement. The presentation order of the two intervention components will be counterbalanced: half of the participants will receive the attention bias task first followed by the interpretation task; the other half will receive the interpretation task first followed by the attention bias task. The intervention is delivered via mobile phone in eight sessions over four weeks (two sessions per week).
  Arms: Gamified-Combined Cognitive Bias Modification
Behavioral: Standard Combined Cognitive Bias Modification — A standard version of the combined cognitive bias modification (CBM-C) intervention, consisting of attention and interpretation bias tasks without gamification features. The attention task is a modified dot-probe paradigm, and the interpretation task involves OCD-related scenarios followed by word-completion exercises. The presentation order of the two intervention components will be counterbalanced: half of the participants will receive the attention bias task first followed by the interpretation task; the other half will receive the interpretation task first followed by the attention bias task. The intervention is delivered via mobile phone in eight sessions over four weeks (two sessions per week).
  Arms: Standart Combined Cognitive Bias Modification
Behavioral: Placebo — A placebo version of the standard CBM-C intervention that retains the same structure and timing but omits all active bias modification elements. The attention task (modified dot-probe) presents probes equally behind threat and neutral stimuli, and the interpretation task includes OCD-related scenarios with word-completion items that lead to neutral outcomes. No manipulations are applied to shift cognitive bias. The presentation order of the two intervention components will be counterbalanced: half of the participants will receive the attention bias task first followed by the interpretation task; the other half will receive the interpretation task first followed by the attention bias task. The intervention is delivered via mobile phone in eight sessions over four weeks (two sessions per week).
  Arms: Placebo Control

SUMMARY:
This randomized controlled trial examines the effects of a mobile-based gamified combined cognitive bias modification (CBM-C) intervention on obsessive-compulsive symptoms, obsessive beliefs, attentional and interpretation biases, depressive symptoms, and psychological distress. The gamified CBM-C condition is compared to a standard mobile-based CBM-C and a placebo control condition. All interventions are delivered via a mobile application. Assessments are conducted at baseline, post-intervention (week 4), and 3-month follow-up.

DETAILED DESCRIPTION:
Cognitive Bias Modification (CBM) is a cognitive intervention that experimentally modifies cognitive biases by using a series of disorder-related stimuli designed to manipulate cognitive processes relevant to psychopathology. There are two major forms of CBM interventions: Cognitive Bias Modification-Attention (CBM-A) and Cognitive Bias Modification-Interpretation (CBM-I). CBM is also a promising treatment for Obsessive- Compulsive Disorder (OCD). In recent years, there has been a growing consensus that there may be causal relations among different cognitive biases ("combined cognitive bias hypothesis"). In line with this hypothesis, it is reasonable to suggest that modification in one section will also have an impact on other biases. There are a few studies testing the effect of Combined CBM (CBM-C) programs on anxiety symptoms, depressive symptoms, and OCD symptoms in subclinical samples with promising results.

In recent years, gamification has also been used in order to increase motivation and participation in experimental tasks that constitute the content of both CBM-A and CBM-I interventions. It is possible to see examples of this method in the field of mental health in general and it is stated that it has the potential to be effective as an intervention on reducing the symptoms of psychiatric disorders. However, there is no study to investigate the effect of gamified CBM in individuals with OCD. Based on these new developments and their positive effects, the aim of the study is to investigate the effect of the gamified CBM-C on reducing the severity of OCD symptoms, obsessive beliefs, interpretation and attentional biases, depressive symptoms, and psychological distress, and increasing motivation and participation in experimental tasks.

The study will be conducted on adult participants primarily diagnosed with OCD according to the DSM-5 criteria by a psychiatrist at Dokuz Eylul University Hospital and referred for outpatient treatment at the same hospital. Participants will be randomly assigned to one of three groups: gamified CBM-C, standard CBM-C, or a placebo control condition. The intervention will be delivered via a mobile phone. Data collection will include self-report assessments and behavioral tasks. Attentional bias will be measured using a dot-probe task with eye-tracking, and interpretation bias will be assessed through a recognition scenario task. Measurements will be taken at baseline, post-intervention (week 4), and at 3-month follow-up.

It is expected that participants in the gamified CBM-C condition will demonstrate greater improvements across clinical symptoms, cognitive biases, and motivational outcomes compared to participants in the standard CBM-C and placebo control groups. To the best of current knowledge, this study will be the first to evaluate the effects of a gamified CBM-C intervention in individuals diagnosed with OCD. Its findings are anticipated to contribute to the development of scalable, accessible, and cost-effective digital interventions for clinical populations with elevated dropout and relapse rates.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Primary diagnosis of obsessive-compulsive disorder (OCD), confirmed by a licensed clinician using the Structured Clinical Interview for DSM-5 (SCID-5)
* No current suicidal ideation or psychotic symptoms
* Access to the internet and a mobile phone
* Stable psychiatric medication use for at least one month prior to enrollment, with no changes in dosage during the 4-week intervention period
* No current neurological or medical condition that would interfere with participation
* Ability to perceive colored visual stimuli (e.g., no color blindness)
* Not currently enrolled in another intervention-based study
* Not receiving any other form of psychological treatment at the time of participation

Exclusion Criteria:

* Presence of active suicidal ideation or psychotic symptoms
* Unstable psychiatric medication use (e.g., recent dose change within the past month or expected change during the intervention period)
* Significant neurological or medical illness that may interfere with participation
* Visual impairments that would prevent accurate perception of colored stimuli (e.g., color blindness)
* Current participation in another clinical trial involving psychological intervention
* Receiving concurrent psychotherapy or other psychological treatments outside of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-04-02 (Estimated); Study Completion 2027-04-02 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale | Baseline, Post-Intervention (Week 4), 3-Month Follow-Up
  This clinician-administered measure is used to assess the severity of obsessive-compulsive symptoms. It includes 19 items in total; however, only the first 10 items are used to calculate the total score. Each item is rated on a 0 to 4 scale, resulting in a total score range of 0 to 40. Higher scores indicate greater symptom severity (worse outcome).The measure is conducted through a semi-structured clinical interview.
Obsessive Beliefs Questionnaire-44 | Baseline, Post-Intervention (Week 4), 3-Month Follow-Up
  This self-report measure is used to assess dysfunctional beliefs commonly associated with obsessive-compulsive symptoms. It consists of 44 items rated on a Likert-type scale ranging from 1 to 7. The total score ranges from 44 to 308. Higher scores indicate that the individual has more maladaptive obsessive-compulsive beliefs (worse outcome).
OC bias index | Baseline, Post-Intervention (Week 4), 3-Month Follow-Up
  Measure of interpretation biases. It is a computerized task that requires participants to read and imagine themselves in 10 OC-relevant test scenarios and 10 non-OC-relevant scenarios with a title and missing letter in the final word of the sentence. Participants are then provided with a recognition rating form where they see the title of only the 10 OC-relevant scenarios in which they had previously imagined themselves. Each title corresponds with four different interpretations: target bias (OC-positive and OC-negative), and foil bias (foil-positive and foil-negative). Participants are asked to rate (on a 4-point scale) each sentence independently in terms of how similar each interpretation option is to the meaning of the scenario they had previously read. Target and Foil Bias Index scores are calculated by subtracting ratings for negative items from ratings for positive items. A positive score indicates that the individual has more OC-positive interpretations (better outcome).
Dot-Probe Task with Eye-Tracking | Baseline, Post-Intervention (Week 4), 3-Month Follow-Up
  A computerized task measuring attention bias using 48 trials combining probe type, position, and image type (neutral vs. OCD-related). Each trial includes a fixation cross (500 ms), a picture pair (1500 ms), and a directional probe replacing one image. Participants respond via keyboard; bias scores are calculated by subtracting response times for probes replacing OCD-related vs. neutral images. More negative bias scores indicate reduced attention to OCD-related stimuli (better outcome). Eye-tracking (Gazepoint HD 150Hz) measures (a) vigilance: first fixation latency and frequency (including direction bias), (b) disengagement: first fixation duration, and (c) sustained attention: total fixation count and duration. Post-assessment reductions in early, frequent, or prolonged fixations on OCD-related stimuli compared to baseline are interpreted as improved attentional control (better outcome).

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | Baseline, Post-Intervention (Week 4), 3-Month Follow-Up
  This clinician-rated measure is used to assess the severity of depressive symptoms. The version used includes 17 items, each rated on a scale of 0 to 2 or 0 to 4, depending on the item. Total scores range from 0 to 52. Higher scores indicate greater severity of depressive symptoms (worse outcome). The assessment is conducted through a structured clinical interview.
Kessler Psychological Distress Scale | Baseline, Post-Intervention (Week 4), 3-Month Follow-Up
  This self-report measure is used to assess general psychological distress based on symptoms of anxiety and depression experienced over the past 30 days. It includes 10 items rated on a 5-point scale from 1 to 5. Total scores range from 10 to 50, with higher scores indicating greater levels of distress (worse outcome).

OTHER OUTCOMES:
Feedback Form Questionnaire | 3-Month Follow-Up
  This self-report form is used to assess participants' perceptions and experiences regarding the intervention they received. It consists of three sections: (1) perceived benefit and impact of the intervention, (2) usability and practicality of the program, and (3) qualitative feedback on helpful and unhelpful aspects of the intervention. The first section includes 4 items rated on a 5-point scale from 0 (not at all) to 4 (very much). The second section consists of 4 items rated on a 5-point scale from 1 (strongly disagree) to 5 (strongly agree). The third section includes open-ended questions that allow participants to elaborate on which elements of the intervention were helpful or not. Additionally, the form includes a categorical question assessing participants' views on session duration and an optional space for further suggestions.

CONTACTS AND LOCATIONS:
Overall Officials: Sıla Derin, PhD, Principal Investigator — Dokuz Eylul University, İzmir, Turkey
Locations (1):
- Dokuz Eylul University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No